CLINICAL TRIAL: NCT02637401
Title: Group Dialectical Behavioural Therapy for Mood Instability Within Bipolar Disorder: An Open Trial
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 1415/002
Record Dates: First submitted 2015-12-17; First posted 2015-12-22 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Therapy group: Dialectical behaviour therapy: a psychological therpay involving 16 group sessions plus approximately 5 individual meetings over 4 months.
  Interventions: Behavioral: Dialectical Behaviour Therapy

INTERVENTIONS:
Behavioral: Dialectical Behaviour Therapy

SUMMARY:
Bipolar Disorders (BD) typically involve repeated episodes of both depression and excessively high mood or irritability (hypomania or mania). BD presents considerable challenges for the individual, his or her supporters, and society more generally. Medication is generally considered to be the mainstay treatment, however a substantial number of individuals with BD continue to experience episodes despite use of medication. Furthermore, ongoing mood instability either outside of episodes, or as the main feature of their BD, is a significant difficulty experienced by many. Whilst studies suggest that certain psychological therapies can be helpful for people experiencing full bipolar episodes, or to reduce risk of future episodes, there are no evidencebased psychological therapies available for individuals experiencing ongoing mood instability. Dialectical Behaviour Therapy (DBT) was developed several decades ago as an approach for people with Borderline Personality Disorder. DBT aims to give individuals who experience rapid and intense shifts in affect skills for managing this. Despite the many similarities in the symptoms experienced by individuals with Borderline Personality Disorder and those with Bipolar Disorder only a small number of studies have tested DBT for BD, and no studies to date have specifically investigated DBT as a means to help individuals with ongoing mood instability. We have developed a version of groupbased DBT that draws upon our own research to adapt standard DBT for this client group (DBTBD).

The group is designed to be delivered efficiently within the U.K. healthcare system whilst meeting the needs of individual participants through use of additional individual sessions and a mobile phone application. The current study investigates how acceptable DBTBD is to clinicians and patients, and whether - for the small number of individuals in the study -changes in symptoms and key ways of thinking and behaving appear to take place across the period of treatment.

ELIGIBILITY:
Inclusion criteria for patient participants are: i) aged 18 or over; i) meets DSMV criteria for Bipolar Spectrum Disorder; iii) current bipolar mood instability (over the past two years numerous periods with hypomanic symptoms that do not meet criteria for a hypomanic episode and numerous periods with depressive symptoms that do not meet criteria for a depressive episode, continuing into the past month); iv) client wishes to engage in psychological therapy that focusses primarily on ongoing mood instability and its consequences.

Exclusion criteria are: i) current substance dependence disorder; ii) currently receiving other psychological therapy; iii) the patient is currently actively suicidal; iv) presenting difficulties that are characteristic of Borderline Personality Disorder rather than Bipolar Disorder and that would be an early treatment target in standard DBT (frequent and serious deliberate selfharm, marked disturbance in ability to form or maintain interpersonal relationships); v) presence of another area of difficulty that the therapist and client believe should be the primary focus of intervention (for example panic disorder with agoraphobia, Post Traumatic Stress Disorder); vi) the information available suggests that the person may present a significant risk to other group members (such as aggression, likelihood of carrying out sexual or other exploitation); vii) the person lacks capacity to consent to treatment or research participation; viii) currently experiencing an episode of mania.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with frequent bipolar mood swings.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Acceptability of the therapy (% completing treatment) | 10 months
Acceptability of the therapy and study procedures | 10 months
  Qualitiative feedback from participants
Feasibility of the study procedures | 10 months
  recruitment rate; feedback from referrers and clincians / researchers

SECONDARY OUTCOMES:
Clinical effectiveness | 15 months
  symptoms, quality of life, recovery status. Analysis focuses upon the sensitvity of these measures to change, and pre-post correlations.
Process measures | 10 months
  self report measures of key psychological processes hypothesised to be changed by therapy. Analysis focuses upon the sensitvity of these measures to change, and pre-post correlations.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data would potentially be shared on Open Repository Exeter (University of Exeter's open data repository)

REFERENCES:
- [Derived] Wright K, Palmer G, Javaid M, Mostazir M, Lynch T. Psychological therapy for mood instability within bipolar spectrum disorder: a single-arm feasibility study of a dialectical behaviour therapy-informed approach. Pilot Feasibility Stud. 2020 Apr 15;6:46. doi: 10.1186/s40814-020-00586-1. eCollection 2020. PMID 32318271